CLINICAL TRIAL: NCT04644172
Title: Improving Thinking in Everyday Life: Pilot Study C
Brief Title: Improving Thinking in Everyday Life After Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gitendra Uswatte, Professor, Department of Psychology, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300002814C
Record Dates: First submitted 2020-11-23; First posted 2020-11-25 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Covid-19; Cognitive Impairment
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Pilot RCT with two arms: Immediate and Delayed Treatment with crossover to experimental intervention after 6-month followup. Delayed group is allowed to receive usual care while awaiting crossover. Testing is done for both groups at pre- and post-treatment and 6-month followup.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): The treatment will have 3 components. The first component, Speed of Processing Training, is a computer game. Participants identify targets on the screen as rapidly as possible. The second component is training following shaping principles on simulated instrumental activities of daily living (IADL), such as making a telephone call or generating a shopping list, in the treatment setting. Shaping involves progressively increasingly the complexity of a task in incremental steps as a participant gains mastery. Frequent, positive feedback is another important aspect of shaping. The third component is a set of psychological techniques that will help participants apply the improvements from the game to carrying out tasks that rely on thinking in their daily
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Instrumental Activities of Daily Living Shaping; Behavioral: Transfer Package from CI Therapy
- Delayed Treatment (Other): Participants in this arm will receive testing on the same schedule as the Immediate Treatment up to six-month followup. Delayed Treatment participants will not receive any treatment from the study during this period but will permitted to receive any healthcare that is available on a clinical basis. After six-month followup, participants in this arm will be crossed over to receive the experimental treatment.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Instrumental Activities of Daily Living Shaping; Behavioral: Transfer Package from CI Therapy; Other: Usual Care

INTERVENTIONS:
Behavioral: Speed of Processing Training — Testing involves trainer-guided practice of computerbased video "games." The "games" require the "player" to identify targets that are presented very briefly. In the first level, the player has to identify a target at the center of the screen. In the second level, the player has to identify targets at the center and edge of the screen simultaneously. In the third level, other objects, which serve as decoys, are added. SOPT is aimed at improving the fluidity of mental processing speed (not psychomotor reaction time) so that trainees can process more complex information over briefer periods of time. The training involves practice with feedback. The trainer teaches some task-specific strategies, offer suggestions, encouragement, and personalized modification of difficulty for enhancing performance. Speed and task difficulty level are tailored to trainee ability, trainees practice blocks of 16 trials with a goal of achieving performance of 10 to 12 correct trials for each training block.
  Other Names: SOPT
Behavioral: Instrumental Activities of Daily Living Shaping — In addition to training on the SOPT software, participants will train on tasks that simulate everyday activities that have important cognitive components (e.g., selecting medicine bottles from a cabinet, measuring ingredients to bake a cake, finding information online). The training will follow shaping principles. Activity periods will be divided into trials of specific length, and the performance of the participant will be measured and graphed to provide the participant with feedback on their performance. Verbal praise will be used to reward a participant for improvements in performance. The difficulty of the task will be increased in small increments as a participant gains mastery. The purpose of this component is to serve as a bridge between the SOPT training, which exercises a basic aspect of cognitiven function, and cognitive function in everyday life, which is embedded in the context of multi-part, and multidimensional tasks.
  Other Names: IADL Shaping
Behavioral: Transfer Package from CI Therapy — Behavioral Contract. At the outset of treatment, the therapist negotiates a contract with the participant and caregiver, if one is available.Daily home diary. During treatment, the participants catalog the ADL and IADL for the part of the day spent outside the laboratory. Daily administration of the Cognitive Task Activity Log (CTAL). The CTAL collects information about attempts by the participant to complete ADL and IADL. Problem Solving. The therapist helps participants to think through any barriers to completing ADL and IADL independently. Home skill assignments during treatment. Participants are assigned on a written check-off sheet 10 specific ADL tasks. Home skill assignments after treatment. Toward the end of treatment, a written individualized post-treatment program is developed containing a list of up to 10 IADL for each day of the week. Post-treatment telephone contacts. Participants are contacted during the 12 month period after treatment to evaluate treatment outcomes.
  Other Names: Transfer Package (TP)
Other: Usual Care — Healthcare that is available for adults with cognitive impairment subsequent to COVID-19 in the community on a clinical basis. This includes commercially available, gamified, computerized cognitive training programs.
  Arms: Delayed Treatment

SUMMARY:
The purpose of this initial study is to evaluate a new form of cognitive rehabilitation therapy for improving your ability to think, particularly how rapidly you process information that you receive from your senses, e.g., sight, hearing, and smell. The study will also test how often and how well you carry out tasks that rely on thinking in your daily life. You will be randomly assigned to receive the new therapy soon or about three months later. In other words, your treatment schedule will be determined by chance. The new therapy involves intensive, repetitive cognitive exercises (up to 3.5hr/day for 10 consecutive weekdays) with rest periods interspersed as needed.

DETAILED DESCRIPTION:
The purpose of this pilot study is to develop and test an intervention for slow processing of sensory input that not only increases the speed of processing but also produces improvement in how much and how well adults with this type of cognitive impairment carry out everyday tasks that rely on cognitive function. The intervention will combine Speed of Processing Training (SOPT) with a modified form of the Transfer Package (TP) from Constraint-Induced Movement therapy (CI therapy). SOPT has been shown to increase speed of processing in a variety of patient populations. The Transfer Package has been shown to produce transfer of gains from the treatment setting to everyday life when combined with training of arm use in the treatment in adults after stroke.

This early phase, randomized controlled trial (RCT) will have two arms: Immediate SOPT+TP (experimental group) and Delayed SOPT+TP (control group). The Immediate SOPT+TP group will receive the experimental intervention immediately after pre-treatment testing, and then be followed for a year. The Delayed SOPT+TP group will receive testing on the same schedule as the Immediate group up to 3-month follow-up. Delayed group participants will be permitted to receive care that is available in the community as part of typical clinical care during this period. After 3-month follow-up testing, Delayed group participants will receive the experimental intervention and then be followed up for a year. Thus, the study design is a RCT with a usual care control group featuring crossover to the experimental intervention for that group at 3 month follow-up.

In the experimental intervention, the length of each treatment session will vary from 2 to 3.5 hours per day, the number of treatment days per week will range from 2 to 5, and the number of weeks of treatment will range from 2 to 10. Accordingly, the interval between testing occasions may change depending on the findings from initial pilot work. Total hours of treatment will not exceed 35. Ranges are given rather than precise values because part of the purpose of this pilot work is to decide, on a preliminary basis, what is the best schedule of delivery. In addition, four follow-up telephone calls will be conducted each week for the first month after the end of treatment. Then, a follow-up telephone call will be placed once a month for up to 11 months. These telephone calls will permit elements of the Transfer Package to be delivered remotely, helping the patient to transition from taking part in treatment to living their daily lives. Each telephone call will last 30 to 60 minutes.

If a caregiver is available, the caregiver will be asked to complete interviews about the participant's progress (see below) and will be invited to support the participant in following the Transfer Package elements of the treatment (see below).

The outcomes that will be assessed are: speed of processing, performance of instrumental activities of daily living (IADL) that place demands on cognitive activity in the laboratory setting, and performance of IADL that place demands on cognitive activity outside the laboratory setting.

The diagram immediately below shows the treatment and testing schedule for the Immediate Treatment group.

Informed Consent Interview → Screening → Pre-treatment Testing → Treatment (2-10 weeks) → Post-treatment testing → up to 4 weekly follow-up phone calls → up to 2 monthly follow-up phone calls → 3-month follow-up testing → up to 9 monthly follow-up calls → 12-month follow-up testing

The diagram immediately below show the treatment and testing schedule for the Delayed Treatment group.

Informed Consent Interview → Screening → Baseline Testing 1 → Usual care (2-10 weeks) → Baseline Testing 2 → 3 months → Pre-treatment Testing → Treatment (2-10 weeks) → Post-treatment testing → up to 4 weekly follow-up phone calls → up to 2 monthly follow-up phone calls → 3-month follow-up testing → up to 9 monthly follow-up calls → 12-month follow-up testing

Repeated measures analysis of variance models with a between-subjects factor will be used to evaluate if statistically significant improvements take place as a result of treatment. The primary comparison will be between the Immediate Treatment and Delayed Treatment groups at post-treatment. The cross-over design permits a another, secondary evaluation of the efficacy of the experimental intervention by comparing the usual care to the SOPT+TP period in the Delayed Treatment group.

ELIGIBILITY:
Inclusion Criteria:

* presence of cognitive impairment due to Covid-19 infection
* mild-to-moderate general cognitive impairment as determined by a Montreal Cognitive Assessment (MOCA) score between 10-25
* at least 3 months after positive status for Covid-19
* 18 years or older
* medically stable
* sufficiently fit, from both a physical and mental health perspective, to take part in study
* adequate sight and hearing to complete UFOV test
* adequate thinking skills, e.g., ability to follow directions, retain information, to complete UFOV and CTAL, as marked by judgement of the screener that the candidate is able to adequately complete the UFOV and CTAL
* reside in the community (as opposed to a hospital or skilled nursing facility)
* able to travel to laboratory on multiple occasions
* caregiver available

Exclusion Criteria:

- cognitive impairment due to a developmental disability, psychiatric disorder, or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Canadian Occupation Performance Measure (COPM) | Change from Day 0 to Day 17
  The COPM is a widely used, transdiagnostic, individualized, structured interview that detects changes over time in a respondent's performance of five, self-selected activities of daily living (ADL). In this case, the instrument will be completed by a family caregiver and only assess instrumental ADL (IADL) with important cognitive components. Performance is rated using 10-point scale that ranges from 1-10 scale points. High scores reflect effective performance. The test score is the mean of the ratings of the five, self-selected IADL.

SECONDARY OUTCOMES:
Improved and New Cognitive Ability (INCA) | Change from Day 0 to Day 17
  The INCA gathers a comprehensive record of participant changes in everyday Instrumental Activities of Daily Living (IADL) with important cognitive components that have been observed since the start of training. These can be reported by the participant (when possible), the caregiver, or other friends and family that have spent time with the participant. The test score is a count; it is the number of new and improved activities with important cognitive components that a participant has been observed to undertake in their daily life since beginning training. The range is 0 to infinite.
Cognitive Task Activity Log (CTAL) How Well Scale | Change from Day 0 to Day 17
  The CTAL quantifies how well and independently participants complete activities of daily living (ADL) and instrumental ADL (IADL) outside the treatment setting. Twenty-two activities with important cognitive components are surveyed; each is rated by the family caregiver using 11-point scales. The How Well Scale is reported here. The range is 0-5 scale points; high scores reflect effective performance of the activities.
Cognitive Task Activity Log (CTAL) Independence Scale | Change from Day 0 to Day 17
  The CTAL quantifies how well and independently participants complete activities of daily living (ADL) and instrumental ADL (IADL) outside the treatment setting. Twenty-two activities with important cognitive components are surveyed; each is rated by the family caregiver using 11 point scales. The Independence Scale is reported. The range is 0-5 scale points; high scores reflect performance of the activities without assistance from others.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Taub, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This is pilot study. A major purpose of this study is simply to develop the intervention. Sharing individual data is premature.

REFERENCES:
- [Derived] Uswatte G, Taub E, Ball K, Mitchell BS, Blake JA, McKay S, Biney F, Iosipchuk O, Hempfling P, Harris E, Dickerson A, Lokken K, Knight AJ, Mark VW, Agnihotri S, Cutter G. Long COVID brain fog treatment: An early-phase randomized controlled trial of constraint-induced cognitive therapy signals go. Rehabil Psychol. 2025 Apr 28:10.1037/rep0000626. doi: 10.1037/rep0000626. Online ahead of print. PMID 40310209